CLINICAL TRIAL: NCT00565084
Title: A Randomized, Placebo-Controlled Single-Dose 3-Period Crossover Study to Assess the Tolerability and Efficacy of Ibuprofen 800 mg in a Walking Model of Osteoarthritis Pain
Brief Title: Tolerability and Efficacy of Ibuprofen 800 mg in a Walking Model of Osteoarthritis Pain (0000-057)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-057; 057; 2007_649
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): Ibuprofen
  Interventions: Drug: ibuprofen
- 2 (Placebo Comparator): Placebo 1
  Interventions: Drug: Placebo
- 3 (Placebo Comparator): Placebo 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibuprofen — Patients will receive 800 mg ibuprofen in one of the three treatment periods.
  Arms: 1
Drug: Placebo — Patients will receive placebo to ibuprofen in two of the three treatment periods.
  Arms: 2; 3

SUMMARY:
The purpose of the study is to see if generic ibuprofen has an effect on osteoarthritis knee pain during a series of timed walks on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* The primary source of pain is the study knee of one lower extremity
* Patient is willing to limit alcohol and caffeine intake
* Aside from osteoarthritis, patient is in generally good health
* Patient is capable of completing protocol specified walks
* Patient is able to understand and complete questionnaires in English
* Patient has previously benefited from the use of either NSAIDs, COX-2 inhibitors, or acetaminophen

Exclusion Criteria:

* Patient has another condition which could interfere with evaluating pain in the knee being tested
* Patient is not able to take a non-steroidal anti-inflammatory drug (NSAID) such as ibuprofen
* Patient has a history or current evidence of stroke, transient ischemic attack, liver disease or cancer
* Patient has a history or current evidence of dizziness, unsteadiness, or falling
* Patient has congestive heart failure, unstable angina or uncontrolled high blood pressure
* Patient has a history of stomach, digestive track, or small intestine surgery
* Patient is unable to complete the study questionnaires in English

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Peeva E, Beals CR, Bolognese JA, Kivitz AJ, Taber L, Harman A, Smugar SS, Moskowitz RW. A walking model to assess the onset of analgesia in osteoarthritis knee pain. Osteoarthritis Cartilage. 2010 May;18(5):646-53. doi: 10.1016/j.joca.2009.12.008. Epub 2010 Feb 6. PMID 20175977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered 16 Mar 2007
  Multicenter, 3 sites
Pre-assignment Details: This study is a single dose, multi-center, randomized, placebo controlled, cross-over study using the Walking Model of Osteoarthritis (OA) knee pain. The efficacy and tolerability of a single dose of Ibuprofen 800 mg in the setting of standardized walks will be compared with placebo.
Groups:
- Placebo-Placebo-Ibuprofen: First single dose placebo; second single dose placebo; single dose ibuprofen 800 mg
- Placebo-Ibuprofen-Placebo: First single dose placebo; single dose ibuprofen 800 mg; second single dose placebo
- Ibuprofen-Placebo-Placebo: Single dose ibuprofen 800 mg; first single dose placebo; second single dose placebo
Period: First Treatment Period
Arm/Group | Placebo-Placebo-Ibuprofen | Placebo-Ibuprofen-Placebo | Ibuprofen-Placebo-Placebo
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0
Period: Second Treatment Period
Arm/Group | Placebo-Placebo-Ibuprofen | Placebo-Ibuprofen-Placebo | Ibuprofen-Placebo-Placebo
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0
Period: Third Treatment Period
Arm/Group | Placebo-Placebo-Ibuprofen | Placebo-Ibuprofen-Placebo | Ibuprofen-Placebo-Placebo
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 60.78 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pain Intensities Measured From the Pre-Treatment Walk (Baseline) at 3 Post-Treatment Walks
Description: Pain intensities(PIs) were measured at pre-dose and 3 post-dose walks (15 Minutes Each Separated by a 45-Minute Rest Interval) on an 11 point scale(0=no pain; 10=worst pain) and averaged for each walk.
  Change from baseline was average of post-dose PIs minus average of pre-dose PI.
Time Frame: All pain intensities measured from the pre-treatment walk and 3 post-treatment walks (within 3 and half hours post dose, 15 minutes each walk separated by a 45-minute rest interval)
Population: This is a crossover study. Total number of participants was 33; every participant had one ibuprofen period and two placebo periods.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Ibuprofen: Single dose ibuprofen 800 mg
- Placebo 1: First Single dose placebo
- Placebo 2: Second Single dose placebo
Arm/Group | Ibuprofen | Placebo 1 | Placebo 2
Number analyzed (Participants) | 33 | 33 | 33
Units on a Scale | 0.24 (0.77) | 0.18 (0.77) | 0.18 (0.77)
Statistical Analysis 1: Comparison: Ibuprofen vs Placebo 1 vs Placebo 2; Primary efficacy endpoint was assessed by an ANOVA model with terms for treatment, period, sequence, and patients within sequence. Efficacy advantage over placebo was assessed via the treatment difference in the least-squares (LS) means (ibuprofen vs. average of the 2 placebo treatments) from the ANOVA model and the 90% confidence interval (CI; one-sided alpha=0.05) of the LS mean difference will be assessed; Test type: Superiority or Other; p = 0.743, ANOVA; Difference in LS Means = 0.06, 90% CI [-0.23 to 0.35]

ADVERSE EVENTS:
Time Frame: From consent to 14 day follow up after all treatment periods was from 16-Mar-2007 to 10-Dec-2007. First study dosing to last dosing period was from 23-Mar-2007 to 03-Dec-2007.
Arm/Group | Placebo-Placebo-Ibuprofen | Placebo-Ibuprofen-Placebo | Ibuprofen-Placebo-Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 1/11
Other Adverse Events (participants affected / at risk) | 3/11 | 3/11 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo-Ibuprofen (N=11) | Placebo-Ibuprofen-Placebo (N=11) | Ibuprofen-Placebo-Placebo (N=11)
Breast Ductal Cancer Infiltrating (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Breast cancer diagnosed prior to randomization, and considered unrelated to study drug therapy by the investigator.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo-Ibuprofen (N=11) | Placebo-Ibuprofen-Placebo (N=11) | Ibuprofen-Placebo-Placebo (N=11)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Boil on Buttock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cold Symptoms (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Track Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hip Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in Joint involving hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in Hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tibia Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Unilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Tingling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.